CLINICAL TRIAL: NCT00417963
Title: The ViVEXX Carotid Revascularization Trial (VIVA) for High Surgical Risk Patients With Extracranial Carotid Artery Stenosis Using the Bard ViVEXX Carotid Stent and Emboshield BareWire Rapid Exchange Embolic Protection System
Brief Title: ViVEXX Carotid Revascularization Trial (VIVA)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: C. R. Bard (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BPV-VX-1502
Record Dates: First submitted 2007-01-02; First posted 2007-01-04 (Estimated); Results first posted 2011-07-20 (Estimated); Last update posted 2017-03-01 (Actual); Status verified 2017-01

CONDITIONS: Carotid Artery Stenosis
Keywords: Carotid; Artery; Stenosis
MeSH Terms: conditions — Carotid Stenosis; Constriction, Pathologic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- stent placement in the carotid artery (Experimental): placement of a bare metal stent for treatment of carotid artery stenosis
  Interventions: Device: Carotid Artery Stenting

INTERVENTIONS:
Device: Carotid Artery Stenting — placement of a bare metal stent at sites of stenosis in the carotid artery
  Other Names: CAS

SUMMARY:
To evaluate the safety and efficacy of the Bard ViVEXX Carotid Stent and Emboshield BareWire Rapid Exchange Embolic Protection System in the treatment of extracranial carotid artery stenosis in patients at high risk for carotid endarterectomy.

DETAILED DESCRIPTION:
Patients with clinically significant stenosis within the common and/or internal carotid artery who are at high risk for carotid endarterectomy and are amenable to percutaneous treatment including embolic protection, balloon angioplasty and the carotid stent placement.

ELIGIBILITY:
Inclusion Criteria:

* The patient has a symptomatic or asymptomatic carotid artery stenosis that meets one of the following criteria:

  * Symptomatic: > than or = to 50% carotid stenosis by angiography and a history of non-disabling stroke, transient ischemic attack (TIA) in the hemisphere supplied by the target vessel within 180 days of the procedure.
  * Asymptomatic: > than or = to 80% carotid stenosis by angiography without neurological symptoms.
* High risk for carotid endarterectomy: anatomical and co-morbid.

Exclusion Criteria:

* History of symptoms of stroke or TIA within 24 hours of the procedure
* Extensive or diffuse atherosclerotic disease
* Severe vascular tortuosity or anatomy that would preclude the safe introduction of the device

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 407 (Actual)
Dates: Start 2005-10; Primary Completion 2009-01 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Rosenfield, MD, Principal Investigator — Massachusetts General Hospital

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment commenced on October 7, 2005 and was completed on November 6, 2007. A total of 486 patients from 34 investigative sites within the United States were enrolled, including 79 in the roll-in cohort and 407 in the pivotal cohort. The Roll-in cohort is intended to provide initial training and verification of procedure technique
Pre-assignment Details: Each site was required to enroll at least one roll-in patient prior to commencing the pivotal phase to demonstrate appropriate training and technique. Each roll-in patient was required to meet the same eligibility criteria and follow the same follow-up schedule as the pivotal cohort. The pivotal cohort represents the intent-to-treat population.
Groups:
- ViVexx Carotid Stent Group: placement of a bare metal stent for treatment of carotid artery stenosis
Period: Overall Study
Arm/Group | ViVexx Carotid Stent Group
Started | 486 (79 participants were enrolled in the roll-in cohort and 407 in the pivotal cohort.)
Completed | 445 (79 subjects completed in the roll-in cohort and 371 in the pivotal cohort.)
Not Completed | 41
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 18
Not completed — Death | 17
Not completed — Study device could not be deployed | 3

BASELINE CHARACTERISTICS:
Arm/Group | ViVexx Carotid Stent Group
Number analyzed (Participants) | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.1 (9.14)
Gender [Count of Participants; unit: Participants]
  Female | 191
  Male | 295
Region of Enrollment [Number; unit: participants]
  United States | 486

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Patients Experiencing Major Adverse Events (MAE)
Description: A composite of major adverse events (MAE) including any death, any stroke and/or myocardial infarction occurring during the first 30 days post-procedure and ipsilateral stroke between 31 and 365 days post procedure.
Time Frame: 365 days from implantation
Population: All patients who were enrolled in the pivotal cohort were analyzed as an intention to treat population.
Measure: Mean (95% Confidence Interval); unit: percentage of participants
Arm/Group | ViVexx Carotid Stent Group
Number analyzed (Participants) | 486
percentage of participants | 6.9 [4.5 to 9.2]

2. Secondary Outcome: Number of Participants Experiencing Target Lesion Revascularization(s) (TLR)
Description: Number of participants experiencing a Target lesion revascularization(s) up to 12 months after implantation
Time Frame: 12 months from implantation
Population: Number of participants experiencing target lesion revascularization up to 12 months from implantation
Measure: Number; unit: Number of participants
Groups:
- Stent Placement in the Carotid Artery: All subjects who received the ViVexx Carotid Stent.
- Roll-in Cohort: Participants enrolled in the roll-in cohort of the study. Roll-in patients were not included in the intention to treat analysis.
- Pivotal Cohort: Participants who were enrolled in the Pivotal cohort. All Pivotal subjects were included in the intention to treat analysis.
Arm/Group | Stent Placement in the Carotid Artery | Roll-in Cohort | Pivotal Cohort
Number analyzed (Participants) | 486 | 79 | 407
Number of participants | 19 | 2 | 17

3. Secondary Outcome: Number of Patients Experiencing Access Site Complications
Description: Access site complications requiring blood transfusion (> 1 unit) or open surgical repair.
Time Frame: 30 days following implantation
Population: Number of participants experiencing access site complications requiring blood transfusion (>1 unit) or open repair.
Measure: Number; unit: Number of participants
Arm/Group | Stent Placement in the Carotid Artery | Roll-in Cohort | Pivotal Cohort
Number analyzed (Participants) | 486 | 79 | 407
Number of participants | 8 | 1 | 7

4. Secondary Outcome: Number of Participants Experiencing Stroke Related Neurologic Deficit
Description: Number of participants experiencing stroke related neurologic deficit persisting at 30 days and attributed to the index procedure.
Time Frame: 30 days from implantation
Population: Number of participants experiencing stroke related neurologic deficit persisting at 30 days and attributed to index procedure.
Measure: Number; unit: number of participants
Arm/Group | Stent Placement in the Carotid Artery | Roll-in Cohort | Pivotal Cohort
Number analyzed (Participants) | 486 | 79 | 407
number of participants | 11 | 1 | 10

5. Secondary Outcome: Number of Participants Experiencing Device Success
Description: Number of participants with successful delivery and deployment of device with <50% residual stenosis.
Time Frame: at time of implantation
Population: Number of participants with successful delivery and deployment of device with <50% residual stenosis.
Measure: Number; unit: number of participants
Arm/Group | Stent Placement in the Carotid Artery
Number analyzed (Participants) | 486
number of participants
  Vivexx stent success | 462
  Emboshield device success | 462

6. Secondary Outcome: Number of Participants Experiencing Lesion Success
Description: number of participants experiencing achievement of <50% final residual diameter stenosis in the stented segment using the VIVEXX Carotid Stent and the Emboshield Embolic Protection System.
Time Frame: at time of implantation
Population: number of participants with lesion success defined as <50% residual stenosis.
Measure: Number; unit: number of participants
Arm/Group | ViVexx Carotid Stent Group
Number analyzed (Participants) | 486
number of participants | 473

7. Secondary Outcome: Number of Participants Experiencing Restenosis
Description: Number of participants experiencing Restenosis following placement of the ViVexx Carotid Stent.
Time Frame: 12 months after implantation
Population: Number of participants experiencing restenosis through 12 months from implantation.
Measure: Number; unit: number of participants
Groups:
- 6 Month Restenosis: Number of participants with restenosis at 6 months from implantation.
Arm/Group | Stent Placement in the Carotid Artery | 6 Month Restenosis
Number analyzed (Participants) | 431 | 366
number of participants | 68 | 43

ADVERSE EVENTS:
Time Frame: Implantation through 12 months
Arm/Group | ViVexx Carotid Stent Group
Serious Adverse Events (participants affected / at risk) | 316/486
Other Adverse Events (participants affected / at risk) | 301/486
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | ViVexx Carotid Stent Group (N=486)
Anaemia (Blood and lymphatic system disorders) | 21
Iron deficiency anaemia (Blood and lymphatic system disorders) | 2
Leukocytosis (Blood and lymphatic system disorders) | 3
Splenomegaly (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 1
Angina pectoris (Cardiac disorders) | 4
Angia unstable (Cardiac disorders) | 1
Aortic valve stenosis (Cardiac disorders) | 1
Arrythmia (Cardiac disorders) | 4
Atrial Figrillation (Cardiac disorders) | 15
Arterioventricular block first degree (Cardiac disorders) | 1
Bradycardia (Cardiac disorders) | 12
Bundle branch block right (Cardiac disorders) | 1
Cardiac Arrest (Cardiac disorders) | 3
Cardiac failure congestive (Cardiac disorders) | 8
Cardiomegaly (Cardiac disorders) | 1
Coronary artery disease (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 8
Palpitations (Cardiac disorders) | 1
Sinus bradycardia (Cardiac disorders) | 6
Tachycardia (Cardiac disorders) | 1
Ventricular extrasystoles (Cardiac disorders) | 2
Ventricular tachycardia (Cardiac disorders) | 4
Atrial septal defect (Congenital, familial and genetic disorders) | 1
Congenital arterial malformation (Congenital, familial and genetic disorders) | 1
Deafness (Ear and labyrinth disorders) | 2
Ear Pain (Ear and labyrinth disorders) | 4
Tinnitus (Ear and labyrinth disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Amaurosis fugax (Eye disorders) | 1
Conjunctival heamorrhage (Eye disorders) | 1
Eye Pain (Eye disorders) | 1
Gaze palsy (Eye disorders) | 2
Halo vision (Eye disorders) | 1
Macular degeneration (Eye disorders) | 2
Orbital oedema (Eye disorders) | 1
Retinal artery embolism (Eye disorders) | 1
Rtinal vein occlusion (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Visual impairment (Eye disorders) | 1
Hypothyrodism (Endocrine disorders) | 4
Inappropriate antidiuretic hormone secretion (Endocrine disorders) | 1
Abdominal hernia (Gastrointestinal disorders) | 1
Abdominal pain (Gastrointestinal disorders) | 4
Abdominal pain upper (Gastrointestinal disorders) | 1
Abdominal tenderness (Gastrointestinal disorders) | 1
Colonic polyp (Gastrointestinal disorders) | 3
onstipation (Gastrointestinal disorders) | 7
Dental caries (Gastrointestinal disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 6
Diverticulum (Gastrointestinal disorders) | 1
Epigastric discomfort (Gastrointestinal disorders) | 1
Gastritis (Gastrointestinal disorders) | 3
Gastrointestinal disorder (Gastrointestinal disorders) | 1
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Hiatus hernia (Gastrointestinal disorders) | 3
Impaired gastric emptying (Gastrointestinal disorders) | 1
Nausea (Gastrointestinal disorders) | 7
Oral disorder (Gastrointestinal disorders) | 1
Stomach discomfort (Gastrointestinal disorders) | 1
Tooth impacted (Gastrointestinal disorders) | 1
Toothache (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Adverse drug reaction (General disorders) | 4
Dyspepsia (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Asthenia (General disorders) | 1
Catheter site haemorrhage (General disorders) | 1
Chest discomfort (General disorders) | 2
chest pain (General disorders) | 12
fatigue (General disorders) | 3
Gait disturbance (General disorders) | 1
Implant site erosion (General disorders) | 1
Infusion site extravasation (General disorders) | 1
Injection site haematoma (General disorders) | 11
Injection site haemorrhage (General disorders) | 1
Injection site pain (General disorders) | 1
mass (General disorders) | 1
Non-cardiac chest pain (General disorders) | 2
Oedema peripheral (General disorders) | 10
Pyrexia (General disorders) | 5
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 3
Hepatic cirrhosis (Hepatobiliary disorders) | 1
Drug hypersensitivity (Immune system disorders) | 2
Acute sinusitis (Infections and infestations) | 1
Adenoviral upper respitaory infections (Infections and infestations) | 1
Bacterial disease carrier (Infections and infestations) | 1
Bronchitis (Infections and infestations) | 4
Cellulitis (Infections and infestations) | 3
Clostridial infection (Infections and infestations) | 1
Clostridium defficile colitis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Herpes zoster (Infections and infestations) | 3
Infection (Infections and infestations) | 2
Labyrinthitis (Infections and infestations) | 1
Otitis externa (Infections and infestations) | 2
Pneumonia (Infections and infestations) | 10
Sinusitis (Infections and infestations) | 3
Skin Candida (Infections and infestations) | 1
Tooth infection (Infections and infestations) | 1
Tracheobronchitis (Infections and infestations) | 1
Upper respiratory tract infection (Infections and infestations) | 3
Urinary tract infection (Infections and infestations) | 14
Urinary tract infection enterococcal (Infections and infestations) | 1
Viral infection (Infections and infestations) | 1
Anaemia postoperative (Injury, poisoning and procedural complications) | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1
Contusion (Injury, poisoning and procedural complications) | 1
fall (Injury, poisoning and procedural complications) | 4
Fibula fracture (Injury, poisoning and procedural complications) | 1
Incisional hernia (Injury, poisoning and procedural complications) | 1
Pelvic Fracture (Injury, poisoning and procedural complications) | 1
Seroma (Injury, poisoning and procedural complications) | 1
Skin laceration (Injury, poisoning and procedural complications) | 3
Spinal compression fracture (Injury, poisoning and procedural complications) | 1
Vascular access complication (Injury, poisoning and procedural complications) | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 2
Wound (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Blood creatine phospokinase MB increased (Investigations) | 1
Blood magnesium decreased (Investigations) | 1
Electrocardiogram QT prolonged (Investigations) | 1
Full blood count decreased (Investigations) | 1
Haemoglobin decreased (Investigations) | 6
Heart rate decreased (Investigations) | 1
Heart rate irregular (Investigations) | 1
NIH stroke scale abnormal (Investigations) | 1
Neurological examination abnormal (Investigations) | 1
Troponin (Investigations) | 1
Troponin increased (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 3
Gout (Metabolism and nutrition disorders) | 2
Hyperglycaemia (Metabolism and nutrition disorders) | 2
Hyperkalaemia (Metabolism and nutrition disorders) | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 2
Hypokalaemia (Metabolism and nutrition disorders) | 3
Hypomagnesaemia (Metabolism and nutrition disorders) | 1
Hyponatraemia (Metabolism and nutrition disorders) | 3
Iron deficiency (Metabolism and nutrition disorders) | 1
Lactic acidosis (Metabolism and nutrition disorders) | 1
Malnutrition (Metabolism and nutrition disorders) | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 3
Arthritis (Musculoskeletal and connective tissue disorders) | 2
Back Pain (Musculoskeletal and connective tissue disorders) | 6
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 5
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1
Musculoskeletal discomfort (Musculoskeletal and connective tissue disorders) | 1
Musculskeletal pain (Musculoskeletal and connective tissue disorders) | 3
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 2
Neck pain (Musculoskeletal and connective tissue disorders) | 5
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 2
Osteopenia (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 3
Arthropathy (Musculoskeletal and connective tissue disorders) | 1
Colon adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Lung neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Skin cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Thyroid neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Aphasia (Nervous system disorders) | 1
Areflexia (Nervous system disorders) | 1
Ataxia (Nervous system disorders) | 1
Basilar artery stenosis (Nervous system disorders) | 1
Burning sensation (Nervous system disorders) | 1
Carotid ARtery Stenosis (Nervous system disorders) | 1
Carpal tunnel syndrome (Nervous system disorders) | 2
Cerebral ischaemia (Nervous system disorders) | 8
Cerebrovascular accident (Nervous system disorders) | 5
cognitive disorder (Nervous system disorders) | 4
convulsion (Nervous system disorders) | 4
Diabetic neuropathy (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 22
Dysarthria (Nervous system disorders) | 2
Embolic stroke (Nervous system disorders) | 2
Facial paresis (Nervous system disorders) | 2
Headache (Nervous system disorders) | 14
Hemianopia (Nervous system disorders) | 1
Hypoaesthesia (Nervous system disorders) | 5
Intracranial haematoma (Nervous system disorders) | 1
Ischaemic stroke (Nervous system disorders) | 1
Loss of consciousness (Nervous system disorders) | 1
Momory impairment (Nervous system disorders) | 2
Motor dysfunction (Nervous system disorders) | 1
Nerve compression (Nervous system disorders) | 1
Neuropathy peripheral (Nervous system disorders) | 2
Parkinson's disease (Nervous system disorders) | 1
Presyncope (Nervous system disorders) | 1
Sensory loss (Nervous system disorders) | 2
Paraesthesia (Nervous system disorders) | 4
Speech disorder (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 7
Syncope vasovagal (Nervous system disorders) | 2
Unresponsive to stimui (Nervous system disorders) | 1
Vertebral artery occlusion (Nervous system disorders) | 1
Agitation (Psychiatric disorders) | 1
Anxiety (Psychiatric disorders) | 4
Confusional state (Psychiatric disorders) | 3
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 4
Mental status changes (Psychiatric disorders) | 1
Azotaemia (Renal and urinary disorders) | 1
Bladder distension (Renal and urinary disorders) | 1
Dysuria (Renal and urinary disorders) | 1
Haematuria (Renal and urinary disorders) | 2
Oliguria (Renal and urinary disorders) | 1
Renal cyst (Renal and urinary disorders) | 1
Renal failure (Renal and urinary disorders) | 11
Renal mass (Renal and urinary disorders) | 1
Urinary incontinence (Renal and urinary disorders) | 1
Urinary retention (Renal and urinary disorders) | 5
Erectile dysfunction (Reproductive system and breast disorders) | 1
Scrotal oedema (Reproductive system and breast disorders) | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 1
Atelectasis (Respiratory, thoracic and mediastinal disorders) | 1
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1
cough (Respiratory, thoracic and mediastinal disorders) | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1
Rales (Respiratory, thoracic and mediastinal disorders) | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 1
Sinus disorder (Respiratory, thoracic and mediastinal disorders) | 1
Sleep apnoea syndrome (Respiratory, thoracic and mediastinal disorders) | 2
Acne (Skin and subcutaneous tissue disorders) | 1
Actinic keratosis (Skin and subcutaneous tissue disorders) | 1
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 3
Drug eruption (Skin and subcutaneous tissue disorders) | 3
Ecchymosis (Skin and subcutaneous tissue disorders) | 2
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 1
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Skin lesion (Skin and subcutaneous tissue disorders) | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1
Systemic lupus erythematosus rash (Skin and subcutaneous tissue disorders) | 1
Aneurysm (Vascular disorders) | 1
Aortic aneurysm (Vascular disorders) | 1
arterial restenosis (Vascular disorders) | 2
Arterial spasm (Vascular disorders) | 9
Arterial stenosis (Vascular disorders) | 1
Arteriovenous fistula (Vascular disorders) | 2
Blood pressure fluctuation (Vascular disorders) | 1
Carotid artery dissection (Vascular disorders) | 1
Haematoma (Vascular disorders) | 2
Haemorrhage (Vascular disorders) | 1
Hypertension (Vascular disorders) | 21
Hypotension (Vascular disorders) | 43
Intermittent claudication (Vascular disorders) | 6
Ischaemia (Vascular disorders) | 1
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1
Hypoaesthesia facial (Vascular disorders) | 1
Orthostatic hypotension (Vascular disorders) | 3
Peripheral arterial occlusive disease (Vascular disorders) | 2
Peripheral vascular disorder (Vascular disorders) | 1
Subclavian artery stenosis (Vascular disorders) | 1
Thrombophlebitis (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | ViVexx Carotid Stent Group (N=486)
Anaemia (Blood and lymphatic system disorders) | 56
Angina pectoris (Cardiac disorders) | 27
Atrial fibrillation (Cardiac disorders) | 28
Bradycardia (Cardiac disorders) | 27
CArdiac failure congestive (Cardiac disorders) | 45
Mycardial infarction (Cardiac disorders) | 43
Pneumonia (Infections and infestations) | 41
Cerebralvascular accident (Nervous system disorders) | 36
Dizziness (Nervous system disorders) | 32
Renal Failure (Renal and urinary disorders) | 39
Hypertension (Vascular disorders) | 43
Hypotension (Vascular disorders) | 107

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days